CLINICAL TRIAL: NCT01684748
Title: Angiotensin II Blockade and Adipose Tissue Inflammation in Obesity
Brief Title: Angiotensin II Blockade and Inflammation in Obesity
Acronym: ARB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: arbfat
Record Dates: First submitted 2012-09-06; First posted 2012-09-13 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Overweight; Obese; Prehypertension; Hypertension
Keywords: angiotensin II; obesity; diabetes
MeSH Terms: conditions — Overweight; Obesity; Prehypertension; Hypertension; Diabetes Mellitus | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olmesartan Medoxomil first, then No Drug (Experimental): During the First Intervention (8 weeks), subjects will be provided with daily 20 mg of olmesartan for the first 2 weeks. Subjects receive additional daily doses of 40 mg olmesartan for the remainder of the study period (6 weeks). The dose remains at 20 mg per day, however, if BP falls below 110/70 during the first 2 weeks. In addition, subjects will continue taking the drug during the 2-week follow-up testing period. Subjects will then proceed to the Washout period (2 weeks). During the Second Intervention (8 weeks), no drug will be administered to the subjects.
  Interventions: Drug: Olmesartan medoxomil
- No Drug first, then Olmesartan Medoxomil (Experimental): During the First Intervention (8 weeks), no drug will be administered to the subjects. Subjects will then proceed to the Washout period (2 weeks). During the Second Intervention (8 weeks), subjects will be provided with daily 20 mg of olmesartan for the first 2 weeks. Subjects then receive daily doses of 40 mg olmesartan for the remainder of the study period (6 weeks). The dose remains at 20 mg per day, however, if BP falls below 110/70 during the first 2 weeks. In addition, subjects will continue taking the drug during the 2-week follow-up testing period.
  Interventions: Drug: Olmesartan medoxomil

INTERVENTIONS:
Drug: Olmesartan medoxomil — Crossover intervention comparing antihypertensive medication to no drug intervention.
  Other Names: Benicar

SUMMARY:
Overweight and obesity, which afflicts ~65% of the U.S. population and more than 1 billion people worldwide, increases the risk of developing hypertension. Activation of the renin angiotensin system (RAS) is an important mechanism by which obesity leads to hypertension. In addition to its vasoconstricting and sodium retaining actions, angiotensin II also has potent pro-inflammatory actions including macrophage infiltration and expression of proinflammatory cytokines in target tissues. Adipose tissue and skeletal muscle appear to be a key sites for the generation of proinflammatory cytokines. Although angiotensin II receptor blockade reduces inflammation in many tissues, the effects on adipose tissue and skeletal muscle in humans are not clear. Importantly, the chronic low grade inflammatory state that accompanies obesity complicates hypertension by contributing to insulin resistance and accelerating cardiovascular disease. Therefore, the general aim of the present proposal will be to determine the influence of angiotensin II receptor blockade on adipose tissue and skeletal muscle inflammation and its relation to improvements in insulin sensitivity, if observed, in obese hypertensive humans. To address these aims, 44 obese (BMI>30 kg/m2) hypertensive (BP>140 systolic and/or 90 diastolic) individuals (age=50-65 years) will be randomized to receive 8 weeks of either the angiotensin II receptor antagonist, olmesartan medoxomil, or no treatment in a crossover manner. Subcutaneous adipose tissue and skeletal muscle biopsies will be obtained and insulin sensitivity (intravenous glucose tolerance tests) will be assessed at baseline and following 8 weeks of each intervention. A two week washout period will separate the interventions.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Weight stable for previous 6 months (+2.0kg)
* Sedentary to recreationally active
* Willing to be randomized to treatment or placebo
* Verbal and written informed consent
* Approved for participation by Medical Director (Jose Rivero, M.D.)

Exclusion Criteria:

* Blood pressure outside stated range
* Diabetes or taking diabetes medications
* Total cholesterol >6.2 mmol/L; triglycerides >4.5 mmol/L
* Past or current ischemic heart disease, stroke, respiratory disease, endocrine or metabolic disease, neurological disease, or hematological-oncological disease
* Evidence of renal insufficiency; GFR< 60 ml/min*
* Medications (including but not limited to antihypertensives, statins or other with anti-inflammatory actions) or antioxidant vitamins or supplements
* Known allergy or hypersensitivity to olmesartan or any of its components
* Pregnant or planning to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P. Davy, Ph.D., Principal Investigator — Virginia Polytechnic Institute and State University

RESULTS

PARTICIPANT FLOW:
Groups:
- Olmesartan Medoxomil First, Then No Drug: During the First Intervention (8 weeks), subjects will be provided with daily 20 mg of olmesartan for the first 2 weeks. Subjects receive additional daily doses of 40 mg olmesartan for the remainder of the study period (6 weeks). The dose remains at 20 mg per day, however, if BP falls below 110/70 during the first 2 weeks. In addition, subjects will continue taking the drug during the 2-week follow-up testing period. Subjects will then proceed to the Washout period (2 weeks). During the Second Intervention (8 weeks), no drug will be administered to the subjects.
  Olmesartan medoxomil
Period: First Intervention - 8 Weeks
Arm/Group | Olmesartan Medoxomil First, Then No Drug | No Drug First, Then Olmesartan Medoxomil
Started | 10 | 10
Completed | 8 | 8
Not Completed | 2 | 2
Period: Second Intervention - 8 Weeks
Arm/Group | Olmesartan Medoxomil First, Then No Drug | No Drug First, Then Olmesartan Medoxomil
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olmesartan Medoxomil First, Then No Drug | No Drug First, Then Olmesartan Medoxomil | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.25 (9.8) | 49.75 (14.2) | 49.5 (11.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Body weight [Mean (Standard Deviation); unit: kg] | 102.3 (20.9) | 90.4 (17.7) | 96.3 (19.7)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 34.5 (7.0) | 31.5 (6.8) | 33.0 (6.9)
Body fat [Mean (Standard Deviation); unit: Percentage of fat] | 43.9 (10.5) | 39.8 (13.5) | 41.8 (12.1)
Total fat mass [Mean (Standard Deviation); unit: kg] | 43.1 (15.1) | 34.6 (14.7) | 38.8 (15.0)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 133.7 (10.1) | 140.6 (12.8) | 137.2 (11.7)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 81.0 (5.1) | 80.1 (7.9) | 80.6 (6.4)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 120.6 (68.5) | 106.8 (50.9) | 113.7 (53.6)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 199.5 (38.2) | 207.8 (20.9) | 203.7 (30.1)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 45.5 (9.8) | 55.1 (29.0) | 50.3 (21.5)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 129.9 (34.9) | 131.3 (22.4) | 130.6 (31.2)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 95.8 (10.8) | 99.1 (13.8) | 97.4 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity by Intravenous Glucose Tolerance Testing (Change Over Time)
Description: Data collected from the intravenous glucose tolerance tests included blood concentrations of glucose and insulin. Glucose was measured immediately on a YSI glucose analyzer and insulin was measured via ELISA colormetric kits once all study samples were collected. To analyze changes in insulin sensitivity, the MINMOD software was used. The MINMOD software uses Bergman's minimal model to determine insulin sensitivity during an intravenous glucose tolerance test. Both glucose and insulin values were inserted at each timepoint collected (33 in total over the 3-hour protocol) and the software was run to generate the insulin sensitivity value at baseline and post-test. This information was then used to calculate the change of insulin sensitivity from baseline to post-testing after each 8-week intervention.
Time Frame: Baseline testing to post-testing after 8-week intervention
Population: Results of insulin sensitivity by intravenous glucose tolerance (IVGTT) testing are reported per intervention (Olmesartan Medoxomil and No drug). Only 10 of the 16 study participants who participated in all or some of the study measurements opted to complete or had sufficient data to analyze for each pre- and post-intervention (4 total) IVGTT.
Measure: Mean (Standard Deviation); unit: mu/L/min
Groups:
- Olmesartan Medoxomil: Subjects will be provided with daily 20 mg of olmesartan for the first 2 weeks during the 8-week intervention. Subjects receive additional daily doses of 40 mg olmesartan for the remainder of the study period. The dose remains at 20 mg per day, however, if BP falls below 110/70 during the first 2 weeks, subjects will continue taking the drug during the 2-week follow-up period.
  Olmesartan medoxomil
- No Drug Intervention: The no-drug intervention (i.e., no placebo is provided) is an 8-week no intervention comparison.
Arm/Group | Olmesartan Medoxomil | No Drug Intervention
Number analyzed (Participants) | 10 | 10
mu/L/min | 0.253 (2.7) | -0.804 (2.2)

2. Other Pre Specified Outcome: Collagen Gene Expression in Skeletal Muscle (Change Over Time)
Description: RNA extraction and quantification were determined using an RNeasy Mini Fibrous Kit and DNase I treatment (Qiagen, Valencia, CA, USA) in accordance to the manufacturer's directions for mRNA extraction. Quantitative real-time polymerase chain reaction (qRT-PCR) measured the expression of collagen III using an ABI PRISM 7900 Sequence Detection System instrument and TaqMan Universal PCR Master Mix according to the manufacturer's instructions (Applied Biosystems, Foster City, CA, USA). Relative gene expression levels were determined using the number of cycles necessary to reach threshold and results were normalized to cyclophilin B RNA levels.
Time Frame: Baseline testing to post-testing after 8-week intervention
Population: Results are reported for the Olmesartan Medoxomil intervention only; there was insufficient RNA yield for the majority of participants during the no drug treatment. Only 7 of the 16 study participants who participated in the study measurements had sufficient data to analyze the pre- and post-intervention skeletal muscle biopsy tissues.
Measure: Mean (Standard Error); unit: Arbitrary unit (AU)
Arm/Group | Olmesartan Medoxomil
Number analyzed (Participants) | 7
Arbitrary unit (AU)
  Pre-Olmesartan medoxomil | 1491 (510)
  Post-Olmesartan medoxomil | 774 (271)

ADVERSE EVENTS:
Arm/Group | Olmesartan Medoxomil | No Drug Intervention
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No